CLINICAL TRIAL: NCT05266833
Title: Slow-Breathing Curriculum for Stress Reduction in High School Students: A Feasibility Randomized Controlled Trial
Brief Title: Breathing for Adolescent Stress Reduction Feasibility RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health and Human Performance Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 101
Record Dates: First submitted 2022-02-10; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Anxiety; Stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Students in the control class received regular class instruction during the 5 weeks. This instruction did not deviate from regular instruction that was provided to all classes, including the intervention classes. During the intervention period, control group students completed the assessments once per week. The control class is considered a treatment-as-usual active control.
- Self-Paced Breathing (Experimental): The self-paced slow diaphragmatic breathing intervention provided guidance for participants to breathe at a slower pace than normal with brief, organic pauses after each inhale and exhale, and with exhales longer than inhales. Participants were guided to breathe at their own pace while following these principles of longer exhales and brief pauses after each inhale/exhale. They were invited to slow their pace when ready, both during each 5-minute session and over the course of the 5 weeks.
  Interventions: Behavioral: Slow diaphragmatic breathing
- Guide-Paced Breathing (Experimental): The guide-paced slow diaphragmatic breathing intervention comprised slow breathing with all exhales twice as long as the inhales; e.g., a 3-second inhale was followed by a 6-second exhale. Participants were instructed to breathe in sync with the guided pace. The breathing pace slowed over the 5 weeks: for weeks 1-2, the breath pattern comprised a 3-second inhale followed by a 6-second exhale; for weeks 3-4, the timing was 4 and 8, respectively; and was 5 and 10 for the last week.
  Interventions: Behavioral: Slow diaphragmatic breathing

INTERVENTIONS:
Behavioral: Slow diaphragmatic breathing — The curriculum was based on three key breathing components that have been shown to reduce stress in adolescents: slow breathing; diaphragmatic breathing; and extended exhale breathing. Slow breathing entails breathing at a pace slower than normal breathing. Diaphragmatic breathing focuses on breaths starting from the diaphragm or abdominal areas, with abdominal, then lung, then chest expansion during the inhale and a slow, gradual, full release of air in the reverse direction on the exhale. Extended exhale breathing comprises breathing with the exhalation duration longer, often twice as long, as the inhalation.
  Two versions of slow diaphragmatic extended exhale breathing were included in this study. For both, participants did the practice while seated comfortably and breathing through the nose, and were guided to increase the inhale and exhale durations over the 5 weeks. Students followed 5-minute videos for each session.
  Arms: Guide-Paced Breathing; Self-Paced Breathing

SUMMARY:
The purpose of this study was to test a simple slow breathing curriculum for reducing stress among high school students. The curriculum was developed by the Health and Human Performance Foundation and implemented for this study at a public high school in Colorado, United States.

DETAILED DESCRIPTION:
Nearly 1 in 3 US adolescents meet the criteria for anxiety, an issue worsened by the COVID-19 pandemic. Untreated adolescent stress and anxiety can adversely affect teenagers' development, education, and physical and mental health. Although stress-management strategies may seem abundant, many are unscalable or inaccessible for today's youth. Slow diaphragmatic breathing reduces stress and anxiety by downregulating the body's stress response, and is a recommended adolescent stress management strategy. Schools are under pressure to support students in reducing stress, yet diaphragmatic breathing practices are rarely used in school settings. The investigators developed and implemented a 5-week curriculum during COVID-era hybrid learning to conduct the first randomized controlled trial of slow diaphragmatic breathing for stress reduction in a US high school setting.

ELIGIBILITY:
Inclusion Criteria: Students were eligible to participate in this study if they:

1. Were enrolled at study start (baseline period) in one of four senior (12th grade) English classes taught by the teacher who was recruited for the study;
2. Accepted participation in the study, including willingness to abide by the randomization process, by signing student assent on the consent form;
3. Had parental permission to participate in the study, indicated by their signing their consent on the consent form.

Exclusion Criteria: Students were excluded from the study and data collection, but not from class, if they:

1. Chose not to participate; or,
2. Did not receive parental permission.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Feasibility - compliance with breathing curriculum | 5 weeks
  Number of participants completing the breathing practices
Feasibility - compliance with effectiveness assessments | 7.5 weeks
  Number of participants completing the STAI and CO2TT assessments
Feasibility - curriculum ease and tolerability | 1-week followup period
  Ease and tolerability of the breathing curriculum was measured as the average ratings on a scale of 0 to 3 (worst to best) of responses about the curriculum's ease, usefulness, and tolerability.
Feasibility - effectiveness assessments ease and tolerability | 1-week followup period
  Ease and tolerability of the preliminary effectiveness assessments was measured as the average ratings on a scale of 0 to 3 (worst to best) of responses about the effectiveness assessments' ease and tolerability.

SECONDARY OUTCOMES:
Change in in-the-moment stress levels from before to after breathing exercises, as measured by the State-Trait Anxiety Inventory, State (STAI-State) Scale, short version. | 5 weeks
  6-item STAI-State, short version scale. Responses are scored from 1 to 4. Final scores range from 6 to 24, with higher scores reflecting higher levels of in-the-moment anxiety.
Change in general stress levels from before to after the 5-week curriculum, as measured by the State-Trait Anxiety Inventory, Trait (STAI-Trait) Scale. | 1.5-week baseline period and 1-week followup period
  20-item STAI-Trait scale. Responses are scored from 1 to 4. Final scores range from 20 to 80, with higher scores reflecting higher levels of general anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya GK Bentley, PhD, Principal Investigator — Health and Human Performance Foundation
Locations (1):
- Aspen High School, Aspen, Colorado, United States

REFERENCES:
- [Derived] Bentley TGK, Seeber C, Hightower E, Mackenzie B, Wilson R, Velazquez A, Cheng A, Arce NN, Lorenz KA. Slow-Breathing Curriculum for Stress Reduction in High School Students: Lessons Learned From a Feasibility Pilot. Front Rehabil Sci. 2022 Jul 1;3:864079. doi: 10.3389/fresc.2022.864079. eCollection 2022. PMID 36189008

DOCUMENTS (1):
  • Informed Consent Form (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT05266833/ICF_000.pdf